CLINICAL TRIAL: NCT06685770
Title: THE EFFECT OF PEROPERATIVE TOTAL INTRAVENOUS ANESTHESIA AND INHALER ANESTHESIA ON POSTOPERATIVE NEUROCGNITIVE DISORDER IN BREAST CANCER SURGERY
Brief Title: EVALUATION OF POSTOPERATIVE NEUROCOGNITIVE IMPAIRMENT
Status: Active, not recruiting | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Munevver Duzgun, Medical Doctor, Haseki Training and Research Hospital
Other Study IDs: HEA-AAR-EK-01
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Neurocognitive Disorder; General Anesthesia; Total Intravenous Anesthesia; Sevoflurane Anaesthesia; Breast Surgery
Keywords: neurocognitive disorder; general anesthesia; mini mental state assessment; mini-cog test
MeSH Terms: conditions — Neurocognitive Disorders | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- total intravenous anesthesia groups: In this study, neurological evaluation tests will be performed before and after surgery for patients who will undergo surgery for breast cancer. All patients will be followed during the perioperative period according to the standards specified in the American Society of Anesthesia guideline. Neurological evaluations will be performed at the 24th hour before surgery, on the day of surgery, and on the 1st, 3rd and 5th days after surgery. Those who underwent total intravenous anesthesia after peroperative anesthesia management will constitute this group. The total amounts of propofol and remifentanil consumed in this group will be recorded.
  Interventions: Other: Mini mental state assessment test; Other: Mini-cog test
- inhaled anesthesia groups: In this study, neurological evaluation tests will be performed before and after surgery for patients who will undergo surgery for breast cancer. All patients will be followed during the perioperative period according to the standards specified in the American Society of Anesthesia guideline. Neurological evaluations will be performed at the 24th hour before surgery, on the day of surgery, and on the 1st, 3rd and 5th days after surgery. Those who received inhaler anesthesia after peroperative anesthesia management will constitute this group. In this group, Minimal alveolar concentration levels of sevoflurane and total amounts of remifentanil will be recorded.
  Interventions: Other: Mini mental state assessment test; Other: Mini-cog test

INTERVENTIONS:
Other: Mini mental state assessment test — Breast cancer is a very common and important disease in the female population around the world. Anesthesia management during surgery for this disease in the postoperative period should be carefully planned. It will be important to examine the neurocognitive effects of anesthesia management in the postoperative period in this patient group. Today, inhaler and total intravenous anesthesia have advantages as well as disadvantages. It would be valuable to examine its neurocognitive effects in this patient group. In this study, the frequently used Mini mental state assessment test and Mini-cog test will be used.With mini mental state assessment, the patient is asked a number of simple questions to evaluate cognitive functions and each question has certain points. Changes in these score levels preoperatively and postoperatively will be compared within each patient. At the end of the study, preoperative and postoperative changes will be compared statistically between the groups.
  Other Names: neurocognitive assessment test
Other: Mini-cog test — Breast cancer is a very common and important disease in the female population around the world. Anesthesia management during surgery for this disease in the postoperative period should be carefully planned. It will be important to examine the neurocognitive effects of anesthesia management in the postoperative period in this patient group. Today, inhaler and total intravenous anesthesia have advantages as well as disadvantages. It would be valuable to examine its neurocognitive effects in this patient group. In this study, the frequently used Mini-cog test will be used.With Mini-cog test, the patient is asked a number of simple questions to evaluate cognitive functions and each question has certain points. Changes in these score levels preoperatively and postoperatively will be compared within each patient. At the end of the study, preoperative and postoperative changes will be compared statistically between the groups.
  Other Names: neurocognitive assessment test

SUMMARY:
In this prospective study, the effects of different anesthesia methods (total intravenous anesthesia and inhaled anesthesia) on neurocognitive function will be examined in patients undergoing breast-conserving surgery without axillary lymph node dissection. Mini-Mental State Examination and Mini-Cog tests will be administered at specific intervals pre and postoperatively. Anesthesia management will follow standard protocols, and the researcher will not intervent in these processes. The relationship between the type of anesthesia and neurocognitive outcomes will be evaluated based on the collected data.

DETAILED DESCRIPTION:
During the preoperative evaluation process, after identifying patients with breast cancer who will undergo breast-conserving surgery and who will not undergo axillary lymph dissection, who meet the inclusion criteria in the study, neurocognitive evaluations of these patients will be performed by the anesthesiologist with the mini-mental state assessment (MMDD) test and Mini-cog test 24 hours before the preoperative period. These two tests will be repeated by the same doctor in the preoperative waiting room on the day of the operation.

From the preoperative waiting room, patients will be taken to the operation room after premedication with 2mg intravenous midazolam. After all patients are monitored with standard American Society of Anesthesia monitoring (heart rate, peripheral saturation, noninvasive artery monitoring) and electro encephalography monitoring (patient state index (PSI)), the initial values will be recorded before surgery. During induction, 1-2mg/kg propofol, 2mcg/kg Fentanyl and 0.8mg/kg rocuronium will be administered and then the patient will be intubated. Patients will be monitored to be normothermic by body temperature monitoring. If peroperative heart rate and noninvasive arterial pressure values increase by more than 20% of the presurgical basal value, remifentanil will be administered as an intravenous infusion between 0.05-2mcg/kg/min to all patients. During the peroperative period, noninvasive arterial pressure values, saturation values, heart rate, Patient state index values, Suppression rates and times, body temperature values will be recorded on the follow up form as values before the operation, at the beginning of the operation, at 30minute intervals from the beginning of the operation, and before and after extubation at the end of the operation. During surgery, peroperative anesthesia management will be determined as the ideal anesthesia method for the patient, as deemed appropriate by the relevant anesthesiologist, and there will be no intervention by the anesthesiologist performing the neurocognitive evaluation.

Heart Rate, saturation, noninvasive arterial pressure values will be recorded upon entry and exit from the postoperative recovery unit. Postoperative pain monitoring will be done with Visual analog scala(VAS), and to patients with a Visual analog scala value above 3, Tramadol 100mg every 6 hours, Nonsteroidal anti-inflammatory 100mg every 6 hours, and paracetamol 1000mg every 6 hours will be given intravenously if necessary. MMDD test and Mini-cog test will be repeated in all patients by the anesthesiologist just before being transferred from the postoperative recovery unit to the ward and at the 24th hour, 3rd day, and 5th day postoperatively.

After all neurocognitive evaluations of the patients are performed at planned intervals for 1 week, which anesthesia method was applied to the patients in the peroperative period will be determined from the anesthesia follow-up sheet and the total time and amount used will be recorded. Patients who underwent total intravenous anesthesia and inhaler anesthesia will be included in the study. Patients whose anesthesia management is changed during the case will be considered excluded from the study. Anesthesia management of patients during the preoperative and peroperative periods will be planned and implemented as deemed appropriate by the anesthesiologist who follows the patient during the surgery, regardless of this planned study. The researcher performing the neurocognitive evaluation will not have any intervention or knowledge in these processes. The reason why this study was planned as a prospective study is that neurocognitive evaluations are performed prospectively. There will be no intervention in the patient's preoperative, peroperative and postoperative anesthesia management.

At the end of the study, the relationship between neurocognitive values and total intravenous anesthesia and inhaled anesthetics will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with early stage breast cancer who will undergo breast-conserving surgery

Exclusion Criteria:

* Patients receiving neoadjuvant radiotherapy and chemotherapy
* Patients who will undergo axillary lymph dissection and total mastectomy
* Asa 4-5 patients
* Patients without voluntary consent
* Patients with previous surgery or vertebrobasilar insufficiency
* Patients with Carotis stenosis
* Patients with a visual analog scale above 4 in the postoperative recovery unit
* Patients in whom cerebral oxygenation decreased by 15% from the beginning in cerebral oximetry monitoring during the perioperative period
* Patients with bleeding that disrupts hemodynamics during follow-up and bleeding greater than 20% of body volume
* Patients with postoperative intensive care unit follow-up
* Patients with a decrease of more than 20% from the baseline systolic value (based on ward monitoring) during follow-up
* Patients with intraoperative ventilation failure, patients with hypercarbia, hypocarbia
* Patients whose Patient State Index value falls below 25, which is sufficient for the depth of anesthesia, during anesthesia induction or maintenance.
* Patients with known neurological, psychiatric, unstable cardiovascular, renal or hepatic system disease
* Patients with Uncontrolled Hypertension
* Patients with greater than 1st degree heart block
* Patients allergic to α2 adrenergic receptor agonist
* Patients who cannot speak and do not know Turkish
* Alcohol and substance addicted patients
* Patients who have used opioids in the last 24 hours
* Patients who developed sepsis during postoperative follow-up
* Patients with a history of recurrent surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients who applied to the general surgery clinic of Haseki Training and Research Hospital due to the diagnosis of early stage breast cancer (stage 1-2) and planned breast-conserving surgery (mass removal only) will be included in this study. Since the neurocognitive status assessment will be made precisely in these patients, diseases and factors affecting the neurological status will be recorded as non-study factors and these patients will be excluded from the study. Preoperative anxiety scores, comorbidities and regular medications of the patients included in the study will also be recorded.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Decrease in Mini Mental State Assessment test | Preoperative 24 hours before, in the preoperative operating room, at the 1st postoperative hour, on the 1st, 3rd, 5th postoperative days.
  Female patients who will undergo breast cancer surgery will be given a mini mental state assessment test at the preoperative 24th hour, before and after surgery, and on the 1st, 3rd, and 5th postoperative days. In this test, the patient's neurocognitive status will be evaluated by asking simple questions that investigate their mental characteristics. Each question has a score and the total score indicates the patient's condition. In these patients, this test will be repeated at regular intervals after surgery and postoperatively and the results will be recorded.High scores on this test indicate good neurological stability, whereas falling is associated with poor neurological status. Changed in the value as a result of this test will be investigated.

SECONDARY OUTCOMES:
Mini-cog test | Preoperative 24 hours before, in the preoperative operating room, at the 1st postoperative hour, on the 1st, 3rd, 5th postoperative days.
  Mini-cog test will be applied to female patients who will undergo breast cancer surgery at the 24th hour before surgery, before and after surgery, and on the 1st, 3rd and 5th days after surgery. In this test, the patient's neurocognitive status will be evaluated by asking simple questions investigating their mental characteristics. Each question has a score and the total score indicates the patient's condition. In these patients, this test will be repeated at regular intervals during and after surgery and the results will be recorded. High scores on this test indicate good neurological stability, whereas falling is associated with poor neurological status.Changed in value as a result of this test will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Oznur Sen, Associate Professor, Study Director — Haseki Training and Research Hospital; Munevver Kayhan, Medical Doctor, Study Chair — Haseki Training and Research Hospital; Esra Kahya Tepe, Medical Resident Doctor, Principal Investigator — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jo YY, Kim JY, Lee JY, Choi CH, Chang YJ, Kwak HJ. The effect of intraoperative dexmedetomidine on acute kidney injury after pediatric congenital heart surgery: A prospective randomized trial. Medicine (Baltimore). 2017 Jul;96(28):e7480. doi: 10.1097/MD.0000000000007480. PMID 28700489
- [Background] Bocskai T, Kovacs M, Szakacs Z, Gede N, Hegyi P, Varga G, Pap I, Toth I, Revesz P, Szanyi I, Nemeth A, Gerlinger I, Karadi K, Lujber L. Is the bispectral index monitoring protective against postoperative cognitive decline? A systematic review with meta-analysis. PLoS One. 2020 Feb 13;15(2):e0229018. doi: 10.1371/journal.pone.0229018. eCollection 2020. PMID 32053678